CLINICAL TRIAL: NCT05707897
Title: A Study to Assess the Food Effect of TS-142 in Healthy Subjects
Brief Title: A Food Effect Study of TS-142 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TS142-304
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-01

CONDITIONS: Effect of Food
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fed condition (Experimental): Period in which subjects receive a single oral dose of TS-142 tablet in fed condition.
  Interventions: Drug: TS-142 10 mg
- Fasted condition (Experimental): Period in which subjects receive a single oral dose of TS-142 tablet in fasted condition.
  Interventions: Drug: TS-142 10 mg

INTERVENTIONS:
Drug: TS-142 10 mg — Single-dose of 10 mg of TS-142

SUMMARY:
This is a study to assess the food effect of TS-142 preliminary market formulation tablet in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male who are aged 18 years or older but less than 40 years at the time of informed consent
2. Body Mass Index (BMI) of 18.5 or more and less than 25.0 at the screening test
3. Subjects who are judged by the investigators as an eligible for the clinical trial participation based on the screening tests and the tests conducted at treatment period 1.

Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. Subjects who are judged to have any disease by the principal investigator or sub-investigator and are not considered healthy
2. Subjects who have any unsuitable medical history for participation in this study, including respiratory, cardiovascular, gastrointestinal, hepatic, renal, urological, endocrinological, metabolic, hematologic, immunologic, dermatological, neurological, or psychiatric diseases
3. Subjects who have any medical histories including sleep-associated symptoms, narcolepsy-like symptoms, suicidal ideation, or suicidal attempts

Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | Predose and up to 24 hours postdose
  Plasma concentration of unchanged form and its metabolite
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Maximum plasma concentration of unchanged form and its metabolite (Cmax)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Time to maximum plasma concentration of unchanged form and its metabolite (tmax)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Area under the plasma concentration-time curve extrapolated to infinity of unchanged form and its metabolite (AUCinf)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of unchanged form and its metabolite (AUC0-last)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Terminal elimination rate constant of unchanged form and its metabolite (λz)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Elimination half-life of unchanged form and its metabolite (t1/2)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Apparent volume of distribution based on the terminal phase of unchanged form (Vz/F)
Pharmacokinetic parameters | Predose and up to 24 hours postdose
  Apparent total body clearance of unchanged form (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No